CLINICAL TRIAL: NCT06263673
Title: Anti-Diabetic Medications to Fight Parkinson's Disease and Lewy Body Dementia
Brief Title: Anti-Diabetic Medications to Fight PD and LBD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jessica R. Wilson, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-008183
Record Dates: First submitted 2024-02-09; First posted 2024-02-16 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Lewy Body Dementia; Parkinson Disease
MeSH Terms: conditions — Lewy Body Disease; Parkinson Disease | interventions — Sitagliptin Phosphate; dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sitagliptin Group (Experimental): Subjects will receive sitagliptin for the approximately 4-week treatment period.
  Interventions: Drug: Sitagliptin
- Dapagliflozin Group (Experimental): Subjects will receive dapagliflozin for the approximately 4-week treatment period.
  Interventions: Drug: Dapagliflozin
- Placebo Group (Placebo Comparator): Subjects will receive placebo for the approximately 4-week treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin — 100 mg once daily, oral
  Other Names: DPP4 inhibitor therapy
  Arms: Sitagliptin Group
Drug: Dapagliflozin — 10 mg once daily, oral
  Other Names: SGLT2 inhibitor therapy
  Arms: Dapagliflozin Group
Drug: Placebo — Once daily, oral. Looks similar to the study drug, but it contains no active ingredient.
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to test the hypothesis that DPP4 inhibitors and SGLT2 inhibitors are well tolerated and have beneficial neurological effects, specifically for Parkinson's disease and Lewy body dementia.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease or Lewy Body Dementia (diagnosis confirmed by neurologist at Mayo Clinic) with stable neurological treatment in the past approximately three months.
* Glucose intolerance or mild diabetes: The American Diabetes Association criteria for pre-diabetes/ glucose intolerance includes fasting glucose 100-125, random glucose 140-199, or hemoglobin A1C 5.7-6.4% and diabetes is > 125 mg/dL, > 200 mg/dL, and 6.5% or greater, respectively (40). It has been previously reported that 50-80% of individuals with Parkinson's disease have abnormal glucose tolerance (17), so this should not limit recruitment.

Exclusion Criteria:

* Use of insulin or other anti-diabetes medications other than metformin.
* Contraindication to taking a DPP4 inhibitor or SGLT2 inhibitor including: allergy, history of angioedema, pancreatitis, active gallbladder disease, renal impairment with EGFR < 45).
* Bleeding disorder, use of anticoagulants, thrombocytopenia, or severe anemia.
* Use of high dose steroids.
* Current systemic chemotherapy.
* Pregnancy or breastfeeding.
* Recent (within 30 days) or recurrent (defined as more than one in the past 12 months) urinary tract infection or yeast infection.
* Other contraindication that would make study participation unsafe or make study related data unable to be interpreted.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-05-07 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2025-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Wilson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Fighting Parkinson's Disease and Lewy Body Dementia with Anti-Diabetic Medications — https://www.mayo.edu/research/clinical-trials/cls-20563911

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 subjects screen failed prior to randomization assignment.
Groups:
- Sitagliptin Group: Subjects received sitagliptin for the approximately 4-week treatment period.
  Sitagliptin: 100 mg once daily, oral
- Dapagliflozin Group: Subjects received dapagliflozin for the approximately 4-week treatment period.
  Dapagliflozin: 10 mg once daily, oral
- Placebo Group: Subjects received placebo for the approximately 4-week treatment period.
  Placebo: Once daily, oral. Looks similar to the study drug, but it contains no active ingredient.
Period: Overall Study
Arm/Group | Sitagliptin Group | Dapagliflozin Group | Placebo Group
Started | 4 | 4 | 5
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin Group | Dapagliflozin Group | Placebo Group | Total
Number analyzed (Participants) | 4 | 4 | 5 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2 | 4
  >=65 years | 3 | 3 | 3 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 5
  Male | 2 | 3 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 5 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 4 | 3 | 5 | 12
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change in Movement Disorder Society- Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Score
Description: The Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) measures the severity and progression of Parkinson's disease. It consists of four subscales that assess various aspects of the disease, including: Non-motor experiences of daily living-Part 1 (13 questions), Motor experiences of daily living-Part 2 (13 questions), Motor examination-Part 3 (33 questions), and Motor complications-Part 4 (6 questions). Each subscale is calculated as a sum of the questions, rated from 0 (normal)-4 (severe). Thus, the subscale score ranges are: Non-motor experiences of daily living-Part 1 (range 0-52), Motor experiences of daily living-Part 2 (range 0-52), Motor examination-Part 3 (range 0-132), and Motor complication-Part 4 (range 0-24) with higher scores indicating more severe Parkinson's Disease.
Time Frame: Baseline, 4 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Sitagliptin Group | Dapagliflozin Group | Placebo Group
Number analyzed (Participants) | 4 | 4 | 4
score on a scale
  MDS-UPDRS score-part 1 | 3.0 [1.0 to 4.0] | -2.5 [-7.0 to 0.0] | -2.5 [-4.0 to -1.0]
  MDS-UPDRS score-part 2 | 1.5 [0.0 to 4.0] | -3.0 [-4.0 to 0.0] | -0.5 [-3.0 to 1.0]
  MDS-UPDRS score-part 3 | -2.0 [-6.0 to 0.0] | -3.0 [-14.0 to 0.0] | 0.0 [0.0 to 2.0]
  MDS-UPDRS score-part 4 | 0.0 [0.0 to 8.0] | 0.0 [-4.0 to 1.0] | 0.0 [-2.0 to 0.0]
Statistical Analysis 1: Comparison: Sitagliptin Group vs Dapagliflozin Group vs Placebo Group; MDS-UPDRS score-part 1; Test type: Superiority; p = 0.008, ANOVA
Statistical Analysis 2: Comparison: Sitagliptin Group vs Dapagliflozin Group vs Placebo Group; MDS-UPDRS score-part 2; Test type: Superiority; p = 0.020, ANOVA
Statistical Analysis 3: Comparison: Sitagliptin Group vs Dapagliflozin Group vs Placebo Group; MDS-UPDRS score-part 3; Test type: Superiority; p = 0.19, ANOVA
Statistical Analysis 4: Comparison: Sitagliptin Group vs Dapagliflozin Group vs Placebo Group; MDS-UPDRS score-part 4; Test type: Superiority; p = 0.33, ANOVA

2. Primary Outcome: Change in Mini Mental State Examination (MMSE) Score
Description: The MMSE consists of 11 questions used by clinicians to check for cognitive impairment. Total scores range from 0 to 30 with lower scores indicating cognitive impairment.
Time Frame: Baseline, 4 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Sitagliptin Group | Dapagliflozin Group | Placebo Group
Number analyzed (Participants) | 4 | 4 | 4
score on a scale | 1.5 [0.0 to 4.0] | 0.5 [-2.0 to 3.0] | 1.5 [-1.0 to 3.0]
Statistical Analysis 1: Comparison: Sitagliptin Group vs Dapagliflozin Group vs Placebo Group; Test type: Superiority; p = 0.67, ANOVA

3. Secondary Outcome: Change in Fasting Glucose
Description: The change in fasting glucose levels (mg/dL) from baseline to 4 weeks.
Time Frame: Baseline, 4 weeks
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Sitagliptin Group | Dapagliflozin Group | Placebo Group
Number analyzed (Participants) | 4 | 4 | 4
mg/dL | -3.5 [-73.0 to 2.0] | -1.0 [-29.0 to 8.0] | -5.0 [-24.0 to 15.0]
Statistical Analysis 1: Comparison: Sitagliptin Group vs Dapagliflozin Group vs Placebo Group; Test type: Superiority; p = 0.65, ANOVA

4. Secondary Outcome: Change in Orthostatic Blood Pressure
Description: Standing average for 15 minutes of three blood pressures collected by an automated oscillometric device (blood pressure cuff) reported in mm Hg
Time Frame: Baseline, 4 weeks
Measure: Median (Full Range); unit: mmHg
Arm/Group | Sitagliptin Group | Dapagliflozin Group | Placebo Group
Number analyzed (Participants) | 4 | 4 | 4
mmHg
  Systolic Blood Pressure | -0.1 [-2.0 to 11.2] | 3.4 [-6.4 to 18.2] | 4.8 [-44.0 to 12.0]
  Diastolic Blood Pressure | -4.6 [-11.2 to 12.0] | 0.0 [-14.0 to 3.8] | 5.2 [-21.0 to 13.4]
Statistical Analysis 1: Comparison: Sitagliptin Group vs Dapagliflozin Group vs Placebo Group; Systolic Blood Pressure; Test type: Superiority; p = 0.67, ANOVA
Statistical Analysis 2: Comparison: Sitagliptin Group vs Dapagliflozin Group vs Placebo Group; Diastolic Blood Pressure; Test type: Superiority; p = 0.91, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent through study completion, approximately 4 weeks.
Description: Adverse event definition used for this study: An untoward or undesirable experience associated with the use of a medical product (i.e. drug, device, biologic) in a patient or research subject.
  At each contact with the subject, the study team sought information on adverse events by specific questioning and if needed, by examination.
Arm/Group | Sitagliptin Group | Dapagliflozin Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT06263673/Prot_SAP_000.pdf